CLINICAL TRIAL: NCT00627809
Title: Phase 4 Study of Application of Intracoronary Low Dose Streptokinase Complementary to Standard Percutaneous Coronary Intervention in Patients With ST Elevation Acute Myocardial Infarction: Effect of Adjunctive Intracoronary Streptokinase on Late Term Left Ventricular Infarct Size and Volumes in Patients With Acute Myocardial Infarction
Brief Title: Effect of Adjunctive Intracoronary Streptokinase on Late Term Left Ventricular Infarct Size and Volumes in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul University, Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-337
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Acute Coronary Syndromes; Acute Myocardial Infarction; Reperfusion Injury
Keywords: coronary microcirculation; acut myocardial infarction; infarct size; streptokinase; reperfusion
MeSH Terms: conditions — Acute Coronary Syndrome; Reperfusion Injury | interventions — Streptokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Following standard primary percutaneous coronary intervention for ST elevation acute myocardial infarction 250.000 U intracoronary Streptokinase will be given
  Interventions: Drug: Streptokinase; Procedure: primary percutaneous coronary intervention
- 2 (Active Comparator): Standard percutaneous coronary intervention for ST elevation myocardial infarction will be performed
  Interventions: Procedure: primary percutaneous coronary intervention

INTERVENTIONS:
Drug: Streptokinase — intracoronary infusion, 250.000 Units
  Other Names: Streptase (Streptokinase)
  Arms: 1
Procedure: primary percutaneous coronary intervention — balloon catheter, stent

SUMMARY:
The investigators hypothesized that complementary intracoronary streptokinase administration to primary percutaneous intervention in patients with acute myocardial infarction may provide limitation infarct size and improvement in left ventricular volumes and function in acute and late phases (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Continuous chest pain that lasted > 30 minutes within the preceding 12 hours
* ST-segment elevation of at least 1 mm in 2 contiguous leads on the ECG
* Infarct related artery (IRA) occlusion (TIMI grade 0) at the angiography

Exclusion Criteria:

* Contraindications to streptokinase, tirofiban, aspirin, clopidogrel, or heparin
* Culprit lesion in saphenous vein graft
* TIMI grade II-III flow in IRA
* Additional epicardial stenosis in the IRA distal to stented segment (significant or insignificant)
* Presence of left bundle branch block
* History of prior MI

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular infarct size by SPECT | at long term (5-6 months)
Left ventricular diastolic volume | at long term (5-6 months)
Left ventricular systolic volume | at long term (5-6 months)
Left ventricular ejection fraction | at long term (5-6 months)

SECONDARY OUTCOMES:
Temporal changes (from baseline to 5 months follow-up) in microvascular perfusion indices (index of microvascular resistance, coronary flow reserve) and in infarct size have been interrogated in only control group. | early phase (at discharge) and late phase (5-6 months)
Reinfarction | from recruitment until the last follow-up at 5-6 months
Major bleeding | from recruitment to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Murat Sezer, Assoc. Prof., Principal Investigator — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology; Sabahattin Umman, Prof., Study Director — Istanbul University,Istanbul Faculty of Medicine, Department of Cardiology; Arif O Cimen, M.D., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology; Emre K Aslanger, M.D., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology; Berrin Umman, Prof., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology; Zehra Bugra, Prof., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology; Isik Adalet, Prof., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Nuclear Medicine; Cuneyt Turkmen, Assoc. Prof., Study Chair — Istanbul University, Istanbul Faculty of Medicine, Department of Nuclear Medicine
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Sezer M, Oflaz H, Goren T, Okcular I, Umman B, Nisanci Y, Bilge AK, Sanli Y, Meric M, Umman S. Intracoronary streptokinase after primary percutaneous coronary intervention. N Engl J Med. 2007 May 3;356(18):1823-34. doi: 10.1056/NEJMoa054374. PMID 17476008